CLINICAL TRIAL: NCT04780880
Title: Incidence and Prognostic Factors for Lower Extremities Injuries in Polish Youth Soccer Academy.
Status: Withdrawn | Type: Observational
Why Stopped: Study halted prior to enrollment due to logistical challenges and failure to recruit eligible athletes from participating soccer academies.
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Other Study IDs: NKBBN/680/2020; NKBBN/680/2020 (Other: Independent Bioethics Committee for Scientific Research)
Record Dates: First submitted 2021-01-18; First posted 2021-03-04 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2024-02

CONDITIONS: Musculoskeletal Diseases; Athletic Injuries
MeSH Terms: conditions — Musculoskeletal Diseases; Athletic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Youth football players: Young footballers aged 10-16 training and playing for a Polish football club.

SUMMARY:
The aim of our study is to obtain data on the occurrence of injuries, their mechanisms and types among children and adolescents from a youth soccer club. In addition, in order to determine the potential risk of injury, the investigators will examine the prognostic factors on the basis of tests assessing the antropometric, anatomical, physical and fitness characteristics.

DETAILED DESCRIPTION:
During the 2020/2023 seasons, participants will be obliged to report injuries to to sports physiotherapists.

Supervision and data collection on injuries will be documented by experienced sports physiotherapists. Using the Injury Record Form, a standardized definition and classification of injuries in line with the International Olympic Committee Consensus describing methods for recording and reporting epidemiological data on injuries and diseases in sport (Bahr et al. 2020). In addition, the data will also come from a physiotherapeutic examination, and in the case of severe injuries (requiring specialist consultation), a medical examination (orthopedic and / or neurological) and imaging tests.

Training and match exhibition (time spent by participants during training units and match games) will be recorded individually for each participant by the coaches of a given team (year). The given data (in minutes) will allow to determine the total time of sports exposure. The participant's missed training and / or competition due to an injury will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* healthy, not reporting health problems on the day of the examination
* active participation in football competitions in the football club
* having a medical permit to participate in football games
* signed consent of the parent / guardian to participate in the study

Exclusion Criteria:

* unable to participate in the study
* restrictions related to full participation in football games and / or training

Ages: 10 Years to 16 Years | Sex: Male
Age Groups: Child
Study Population: Young male footballers (U10-U16) training and competing in a Polish football club.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
The incidence of sports-related injuries in youth athletics | Injury incidence rates were calculated per 1000 hours of play over the 12-month prospective follow-up
  Injury incidence rates were calculated per 1000 player hours (matches and training) According to a consensus statement on injury definitions and data collection procedures in soccer studies;
The incidence of recurrent sports-related injuries | Recurrent injuries incidence rates were calculated per 1000 hours of play over the 12-month prospective follow-up
  According to a consensus statement on injury definitions and data collection procedures in soccer studies;

SECONDARY OUTCOMES:
Injury severity | Injury severity were calculated per days of rehabilitation over the 12-month prospective follow-up
  Time loss in days (days unable to train)
Injuries according to location | Description of the number of injuries according to location of the injury on the body over the 12-month prospective follow-up
  Location of the injury on the body
Injuries according to type of the injury | Description of injuries according to the type of the injury over the 12-month prospective follow-up
  Type of the injured structure
Muscle flexibility and range of joint motion | over the 12-month prospective follow-up
  Muscle flexibility, range of joint mobility (degrees as measured by a goniometer)
Peak Height Velocity | over the 12-month prospective follow-up
  Peak Height Velocity (PHV) calculated using the 'maturity offset' value (report as "PHV years")
Y-Balance Test | over the 12-month prospective follow-up
  Dynamic Balance of the lower extremities (record as reach distance in centimeters "cm" and normalized reach distance in percentages "%")
Counter Movement Jump, Broad Jump and Single Leg Hop for Distance | over the 12-month prospective follow-up
  Power of the lower limbs measured as distance in single-leg and double-leg jump tasks (record as distance in centimeters "cm")
Functional Movement Screen (FMS) | over the 12-month prospective follow-up
  The Functional Movement Screen (FMS) is a screening tool used to identify limitations or asymmetries in movement patterns. FMS consists of 7 movement tasks (deep squat, lunges, hurdle steps, a push-up, straight-leg raises, shoulder mobility, and rotary stability). Each task will be visually assessed by an experienced physiotherapist and marked on a 4-point scale (0-3, worst-best). The total maximum score that can be obtained is 21 points.
Kinematic analysis of the single-leg movement tasks | over the 12-month prospective follow-up
  Kinematic analysis of the single-leg movement tasks (single-leg squat, single-leg landing) - 2D video analysis - record as degrees of motion of the joints

CONTACTS AND LOCATIONS:
Overall Officials: Bartosz Wilczyński, Principal Investigator — Department of Immunobiology and Environment Microbiology, Medical University of Gdańsk
Locations (1):
- Department of Immunobiology and Environment Microbiology, Medical University of Gdańsk, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lu XL, Zhang SH, Cui ZZ. [Care of severe aplastic anemia treated with immunosuppressive drugs]. Zhonghua Hu Li Za Zhi. 1995 Mar 5;30(3):148-50. No abstract available. Chinese. PMID 7664395
- [Background] Rotbart HA. Enteroviral infections of the central nervous system. Clin Infect Dis. 1995 Apr;20(4):971-81. doi: 10.1093/clinids/20.4.971. PMID 7795102